CLINICAL TRIAL: NCT06557122
Title: A Randomized Controlled Clinical Trial Evaluating the Efficacy of a Unique Advanced Bioengineered Skin Substitute With Standard of Care Versus an Active Comparator With Standard of Care in the Treatment of Non-Healing Diabetic Foot Ulcers
Brief Title: Clinical Study to Compare Two Skin Substitute Categories for Their Effectiveness to Treat Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Encoll Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENC-HEL-DFU-02
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SOC and Advanced Bioengineered Skin Substitute (Other): The SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM boot), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and wound care covering with Helicoll® applied weekly or as needed followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous, second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Dynaflex™ or equivalent).
  Interventions: Device: SOC and Advanced Bioengineered Skin Substitute
- SOC and Active Comparator (Other): The SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM boot), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and wound care covering with Epifix® or Grafix® followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous, second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Dynaflex™ or equivalent).
  Interventions: Other: SOC and Active Comparator

INTERVENTIONS:
Device: SOC and Advanced Bioengineered Skin Substitute — SOC primary dressing with Helicoll®
  Arms: SOC and Advanced Bioengineered Skin Substitute
Other: SOC and Active Comparator — SOC primary dressing with Epifix® or Grafix®
  Arms: SOC and Active Comparator

SUMMARY:
The purpose of this clinical evaluation is to collect patient outcome data on a commercially available 510K FDA cleared advanced skin substitute. The commercially available product is Helicoll® Advanced Skin Substitute.

In this trial two groups of subjects with Wagner 1 diabetic foot ulcers (DFUs), will receive standard of care (SOC) treatment for their condition. Half of the patients will have their SOC treatment with Epifix® or Grafix® and the other half will receive a 510K FDA cleared Helicoll® Advanced Skin Substitute as the primary treatment. The primary endpoint is the percentage wound area reduction of the target ulcer. Secondary endpoints include the proportion of subjects that obtain complete closure over the 5-week treatment period, the time to achieve complete wound closure of the target ulcer by the end of 5 weeks, and mean number of IP applications.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older.
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At randomization, subjects must have a target diabetic foot ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 10.0 cm2 measured post debridement using a ruler to measure wound area.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be full thickness on the foot or ankle that does not probe to bone.
7. Adequate circulation to the affected foot as documented by any of the following methods performed within 3 months of the first screening visit:

   1. TCOM ≥30 mmHg
   2. ABI between 0.7 and 1.3
   3. PVR: Biphasic
   4. TBI ˃0.6
   5. As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle of the target extremity.
8. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. The subject must consent to using the prescribed off-loading method for the duration of the study.
10. The subject must agree to attend the twice-weekly/weekly study visits required by the protocol.
11. The subject must be willing and able to participate in the informed consent process.
12. Patients must have read and signed the IRB approved ICF before screening procedures are undertaken.

Exclusion Criteria:

1. A subject known to have a life expectancy of < 6 months.
2. If the target ulcer is infected or if there is cellulitis in the surrounding skin.
3. Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
4. A subject has an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
5. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy.
6. Topical application of steroids to the ulcer surface within one month of initial screening.
7. A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
8. A subject with a glycated hemoglobin (HbA1c) greater than or equal to 13% taken at or within 3 months of the initial screening visit.
9. A subject with a serum creatinine ≥ 3.0mg/dL within 6 months of the initial screening visit.
10. A subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer.
11. Women who are pregnant or considering becoming pregnant within the next 6 months.
12. A subject with end stage renal disease requiring dialysis.
13. A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
14. A subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments.
15. A subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit.
16. A subject who has a sensitivity to bovine (cattle) or ovine (sheep) material.
17. A subject that is allergic to aminoglycoside antibiotics (gentamycin, tobramycin, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clemente Clinical Research, Los Angeles, California
  - Doctors Research Network, South Miami, Florida
  - Foot and Ankle Specialists of the Mid-Atlantic, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOC and Advanced Bioengineered Skin Substitute | SOC and Active Comparator
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per-Protocol (PP) Population (All Randomized Subjects)
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC and Advanced Bioengineered Skin Substitute | SOC and Active Comparator | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.03) | 61.1 (12.29) | 60.8 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 10 | 12 | 22
  Race/Ethnicity: African American | 1 | 0 | 1
  Race/Ethnicity: Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.5 (5.24) | 29.8 (10.61) | 31.2 (7.93)
Smoker [Count of Participants; unit: Participants]
  Current | 0 | 1 | 1
  Former | 4 | 5 | 9
  Never smoked | 8 | 6 | 14
HbA1c [Mean (Standard Deviation); unit: Percentage] | 7.5 (2.38) | 7.6 (1.69) | 7.6 (2.04)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.08 (0.24) | 0.93 (0.35) | 1.01 (0.30)
Years of DFUs [Mean (Standard Deviation); unit: years] | 5.9 (12.98) | 4.9 (16.45) | 5.4 (14.72)
Prior DFU count [Mean (Standard Deviation); unit: Count of Ulcer] | 3.8 (4.86) | 3.9 (8.25) | 3.9 (6.56)
Other concurrent DFUs (at screening) [Count of Participants; unit: Participants]
  0 | 9 | 10 | 19
  1 | 2 | 0 | 2
  2 | 1 | 2 | 3
History DFU recurrence [Count of Participants; unit: Participants] | 6 | 4 | 10
Amputations, Minor [Count of Participants; unit: Participants]
  0 | 9 | 6 | 15
  1 | 1 | 1 | 2
  2 | 1 | 5 | 6
  5 | 1 | 0 | 1
Major amputations [Count of Participants; unit: Participants] | 0 | 1 | 1
Foot deformities [Count of Participants; unit: Participants]
  Charcot (stable) | 1 | 2 | 3
  Plantar arthrodesis | 0 | 1 | 1
  Ankle tarsal tunnel | 1 | 0 | 1
  No deformities | 10 | 9 | 19
Wound area [Mean (Standard Deviation); unit: cm2] | 2.3 (2.13) | 2.4 (1.77) | 2.35 (1.95)
Wound age [Mean (Standard Deviation); unit: Weeks] | 16.5 (13.63) | 23.8 (12.4) | 20.2 (13.02)
Vertical location [Count of Participants; unit: Participants]
  Plantar | 12 | 11 | 23
  Dorsal | 0 | 1 | 1
DFU position [Count of Participants; unit: Participants]
  Medial | 8 | 7 | 15
  Lateral | 4 | 5 | 9
Anatomical location [Count of Participants; unit: Participants]
  Toe | 3 | 4 | 7
  Forefoot | 5 | 6 | 11
  Midfoot | 4 | 1 | 5
  Heel | 0 | 1 | 1
History offloading type [Count of Participants; unit: Participants]
  No offloading | 1 | 3 | 4
  CAM boot | 7 | 5 | 12
  Surgical shoe | 4 | 4 | 8
Number of sharp debridements [Mean (Standard Deviation); unit: Sharp debridements] | 3.5 (1.45) | 3.8 (0.94) | 3.7 (1.2)
Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants] | 0 | 1 | 1
Hypertension [Count of Participants; unit: Participants] | 11 | 6 | 17
Peripheral Arterial Disease/Peripheral Vascular Disease (PAD/PVD) [Count of Participants; unit: Participants] | 1 | 0 | 1
Chronic Heart Failure (CHF) [Count of Participants; unit: Participants] | 2 | 0 | 2
Leg edema [Count of Participants; unit: Participants] | 1 | 0 | 1
Restricted mobility [Count of Participants; unit: Participants] — Any subject who uses a walker, wheelchair, crutches or canes, and/or has an inability to move freely because of a physical or mental disability, handicap or restriction
  Participants | 0 | 0 | 0
Venous disease [Count of Participants; unit: Participants] | 0 | 0 | 0
Peripheral neuropathy [Count of Participants; unit: Participants] | 8 | 12 | 20
Any psychiatric condition [Count of Participants; unit: Participants] | 2 | 3 | 5
Comorbidity count [Mean (Standard Deviation); unit: Comorbidities] | 7.1 (4.06) | 6.9 (4.06) | 7 (4.06)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wound Area Reduction
Description: Average Percentage of Wound Area Reduction from Treatment Visit 1 to Treatment Visit 4 measured manually with digital photography
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Wound Area Reduction
Arm/Group | SOC and Advanced Bioengineered Skin Substitute | SOC and Active Comparator
Number analyzed (Participants) | 12 | 12
Percentage of Wound Area Reduction | 83.9 (24.93) | 71.3 (36.80)

2. Secondary Outcome: Number of Participants With Repeated Applications
Description: Number of Participants with repeated applications of the Advanced Skin Substitute used to obtain wound closure
Time Frame: 4 weeks
Population: Healed wounds only
Measure: Number; unit: participants
Arm/Group | SOC and Advanced Bioengineered Skin Substitute | SOC and Active Comparator
Number analyzed (Participants) | 6 | 3
participants
  1 Repeated Application | 1 | 0
  2 Repeated Applications | 1 | 1
  4 Repeated Applications | 4 | 2

3. Secondary Outcome: Proportion of Complete Closure
Description: The proportion of subjects that obtain complete closure over the 5-week treatment period
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Advanced Bioengineered Skin Substitute | SOC and Active Comparator
Number analyzed (Participants) | 12 | 12
Participants | 6 | 3

4. Secondary Outcome: Time to Achieve Complete Wound Closure
Description: The time to achieve complete wound closure of the target ulcer by the end of 5 weeks
Time Frame: 5 weeks
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | SOC and Advanced Bioengineered Skin Substitute | SOC and Active Comparator
Number analyzed (Participants) | 12 | 12
Days | 28.3 [27.8 to 28.9] | 26.8 [24.3 to 29.3]

5. Other Pre Specified Outcome: Safety Analysis for Treatment Emergent Adverse Events
Description: The number and type of Treatment Emergent Adverse Events
Time Frame: 5 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: An AE is defined as any unfavorable or unintended sign, symptom or disease that occurs or is reported by the subject to have occurred, or a worsening of a pre-existing condition related to the procedure or medical treatment (device/drug) used.
  AEs will be defined as those events that occur after the first study treatment is applied at TV1, through the final study visit.
Arm/Group | SOC and Advanced Bioengineered Skin Substitute | SOC and Active Comparator
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall not independently publish, publicly disclose, present or discuss any results or information pertaining to study conducted under the mutual agreement until such a multi-center publication is released under Sponsor's direction.

DOCUMENTS (2):
  • Study Protocol (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT06557122/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT06557122/SAP_002.pdf